CLINICAL TRIAL: NCT01596790
Title: Assessment by EPISPOT of Circulating Tumor Cells as an Early Predictive Marker of Response to Chemotherapy and Targeted Therapy in Patients With Metastatic Colorectal Cancer in First Line of Treatment
Brief Title: COLOSPOT Study : Assessment by EPISPOT of Circulating Tumor Cells in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: National Cancer Institute, France (Other Government); Direction Générale de l'Offre de Soins (Other Government); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 8748; ID-RCB 2011-A01130-41 (Other: Afssaps)
Record Dates: First submitted 2012-05-04; First posted 2012-05-11 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Bevacizumab; Circulating tumor cells; Treatment efficiency
MeSH Terms: conditions — Colorectal Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CTC assay (Other): Detection & characterization of viable CTC in the peripheral blood.
  Interventions: Other: Blood analysis by EPISPOT and Cellsearch

INTERVENTIONS:
Other: Blood analysis by EPISPOT and Cellsearch — For each patient, we will perform a counting of CTC before chemotherapy and then at different time points after chemotherapy, using both technologies: EPISPOT and CellSearch®.For the EPISPOT, we will need 15 mL of peripheral blood on EDTA tubes. For each patient, five blood samples will be done: D0, D14, D28, D42 and D56. These different time points will help us to determine when the best moment is for the evaluation of the CTC with this technology.For the CellSearch®, we will need 10 mL of peripheral blood on a specific CellSave tube. Only two samples will be perform: D0 and D28 because Cohen et al. (2008) reported that the best appropriated moment to appreciate the CTC progression is between 3 and 5 weeks after the initiation of the treatment.

SUMMARY:
Treatment of metastatic colorectal cancer needs chemotherapy in most of the cases. During these last years, many new chemotherapies and targeted therapies have been developed improving significantly the overall survival of patients. However, the choice of the therapeutic sequences becomes difficult due to the lack of validated predictive biomarkers of their efficiency. Indeed, only the mutation of the k-ras oncogene is a predictive factor of non-efficacy of the anti-EGFR antibodies. It is thus crucial to identify new biomarkers to propose the best personalized 1rst line therapeutic sequence. One idea would be to enumerate and characterize the circulating tumor cells (CTC) which, as it has been described in a recent study realized by Cohen et al. in patients with metastatic colorectal cancer, would give us an early evaluation of the therapeutic efficiency. In this context, the investigators have developed an innovative technology, the EPISPOT assay (patent of the University Medical Center of Montpellier), that allows the detection & characterization of viable CTC in the peripheral blood. The EPISPOT technology has been already evaluated in the breast and prostate cancer. Thus, the investigators would like to perform a prospective study on a cohort of patients with metastatic colorectal cancer to confirm, with this technology, the predictive value of CTC count for the efficacy of the treatment.

DETAILED DESCRIPTION:
In the aim to study a homogeneous cohort of patients, the investigators will only recruit patients in first line of treatment and treated by 5-FU (IV), IRINOTECAN et BEVACIZUMAB combination.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Colon or rectum adenocarcinoma (based on the histology)
* Visceral metastases (synchronous and/or metachronous)
* Metastatic disease measurable with the RECIST 1.1 criteria
* WHO performance status 0, 1 or 2
* Life expectancy>3 months when starting the treatment
* Chemotherapy in metastatic 1rst line combining a protocol of conventional chemotherapy combining 5-FU and IRINOTECAN (FOLFIRI, XELIRI) associated with bevacizumab
* Follow-up of at least one year
* Collection of the written consent
* Social security affiliation

Exclusion Criteria:

* 2nd line chemotherapy and beyond
* History of other cancers considered not cured
* Active and progressive infection or other serious disease that may not allow the patient to receive the treatment
* refusal to participate
* Patient unable to express his consent
* Pregnant women
* Patient unable to be followed-up for at least one year
* Current participation to another clinical trial
* Patients under guardianship
* Vulnerable people protected by the law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Predictive value of the CTC on the Progression Free Survival | Duration study 3 years
  The primary outcome aims to evaluate the predictive value of the early progression of the CTC performed with the EPISPOT assay on the PFS in a cohort of patients treated with 5-FU, IRNOTECAN et AVASTIN (FOLFIRI or XELIRI-AVASTIN) in 1rst line of metastatic colorectal cancer. The progression disease is assessed based on imagery techniques.

SECONDARY OUTCOMES:
Prognostic value of the CTC detected by EPISPOT | Duration study 3 years
  For the EPISPOT assay, 15 mL of peripheral blood will be collected on EDTA tubes. For each patient, 5 blood samples will be collected: at D0, D14, D28, D42 and D56.
Predictive value of the CTC on the overall survival | Duration study 3 years
  The overall survival will be defined as the time between the beginning of the chemotherapy and death.
VEGF expressions by the CTC | Duration study 3 years
  To evaluate the VEGF expression by the CTC with both technologies, the EPISPOT and the CellSearch®.
Comparison of the results with the CellSearch system vs EPISPOT | Duration study 3 years
  For the Cellsearch assay, 10 mL of peripheral blood will be collected on specific tubes. Only 2 samples will be performed: at D0 and D28.
  The Cellsearch and EPISPOT techniques will be performed in parallel and then compared.

CONTACTS AND LOCATIONS:
Overall Officials: Panabieres Catherine, PhD, Study Director — UH Montpellier
Locations (1):
- Medical Oncology, CHU St Eloi, Montpellier, France

REFERENCES:
- [Derived] Cayrefourcq L, Thomas F, Mazard T, Assenat E, Assou S, Alix-Panabieres C. Selective treatment pressure in colon cancer drives the molecular profile of resistant circulating tumor cell clones. Mol Cancer. 2021 Feb 8;20(1):30. doi: 10.1186/s12943-021-01326-6. PMID 33557844